CLINICAL TRIAL: NCT00917267
Title: A Comparator-Controlled Study to Examine the Effects of Exenatide Once-Weekly Injection on Glucose Control (HbA1c) and Safety in Asian Subjects With Type 2 Diabetes Mellitus Managed With Oral Antidiabetic Medications
Brief Title: A Study to Examine the Effects of Exenatide Once-Weekly Injection on Glucose Control and Safety in Asian Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H8O-MC-GWCK
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Results first posted 2012-12-31 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide; once weekly; Byetta; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: exenatide once weekly
- 2 (Active Comparator)
  Interventions: Drug: exenatide twice daily

INTERVENTIONS:
Drug: exenatide once weekly — 2.0mg subcutaneous injection, once a week
  Arms: 1
Drug: exenatide twice daily — 5mcg subcutaneous injection twice a day (4 weeks), 10mcg subcutaneous injection twice a day (22 weeks)
  Other Names: Byetta
  Arms: 2

SUMMARY:
Previous studies have suggested that a once-weekly formulation of exenatide may provide sustained glycemic control. These previous studies of exenatide once weekly have been conducted in non-Asian populations, so this study has been developed to support the local regulatory requirements of China, Korea, Japan, India, and Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with type 2 diabetes.
* Have suboptimal glycemic control as evidenced by an HbA1c between 7.1% and 11.0% inclusive.
* Have a body mass index (BMI) of >21 kg/m2 and <35 kg/m2, inclusive.
* Have a history of stable body weight (not varying by >5% for at least 90 days prior to study start).
* Have been treated with a stable dose regimen of Met, SU, TZD, Met plus SU, Met plus TZD, or SU plus TZD for at least 90 days prior to study start.

Exclusion Criteria:

* Have any contraindication for the OAD(s) that they use.
* Have a known allergy or hypersensitivity to exenatide BID, exenatide QW, or excipients contained in these agents.
* Have received chronic >14 consecutive days) systemic glucocorticoid therapy by oral, intravenous (IV), or intramuscular (IM) route or intra-articular steroid injection within 4 weeks prior to study start or are regularly treated with potent, inhaled steroids that are known to have a high rate of systemic absorption.
* Have been treated with drugs that promote weight loss (for example, GLP-1 analogue, orlistat, sibutramine, phenylpropanolamine, or similar over-the-counter medications) within 90 days of study start.
* Have been treated for >2 weeks with any of the following excluded medications within 90 days prior to study start:

  * Insulin
  * Dipeptidyl peptidase (DPP)-4 inhibitors (for example, sitagliptin or vildagliptin)
  * Pramlintide acetate
  * Drugs that directly affect gastrointestinal motility, including, but not limited to: Reglan® (metoclopramide), Propulsid® (cisapride), and chronic macrolide antibiotics.
* Have had prior exposure to exenatide
* Have previously completed or withdrawn from this study or any other study investigating exenatide BID or QW.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Are currently enrolled in any other clinical study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 691 (Actual)
Dates: Start 2009-07; Primary Completion 2010-09 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer Officer, MD, Study Director — Eli Lilly and Company
Locations (42):
- China (5):
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Chongqin
  - Research Site, Guangzhou
  - Research Site, Shanghai
- India (12):
  - Research Site, Ahmedabad
  - Research Site, Aligarh
  - Research Site, Bangalore
  - Research Site, Ghaziabad
  - Research Site, Hyderabaad
  - Research Site, Indore
  - Research Site, Kolkata
  - Research Site, Mumbai
  - Research Site, Pune
  - Research Site, Trivandrum
  - Research Site, Uttar Pradesh
  - Research Site, Varanasi
- Japan (16):
  - Research Site, Ageo
  - Research Site, Chiyoda-ku
  - Research Site, Izumisano
  - Research Site, Kashiwara
  - Research Site, Kitaazumi-gun
  - Research Site, Kumamoto
  - Research Site, Kurume
  - Research Site, Matsumoto
  - Research Site, Matsuyama
  - Research Site, Miyazaki
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Ōta-ku
  - Research Site, Shinjuku-ku
  - Research Site, Takatsuki
  - Research Site, Yokohama
- South Korea (3):
  - Research Site, Bucheon-si
  - Research Site, Daegu
  - Research Site, Seoul
- Taiwan (6):
  - Research Site, Changhua
  - Research Site, Chiayi City
  - Research Site, Kaohsiung City
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District

REFERENCES:
- [Derived] Onishi Y, Koshiyama H, Imaoka T, Haber H, Scism-Bacon J, Boardman MK. Safety of exenatide once weekly for 52 weeks in Japanese patients with type 2 diabetes mellitus. J Diabetes Investig. 2013 Mar 18;4(2):182-9. doi: 10.1111/jdi.12000. Epub 2012 Oct 22. PMID 24843650
- [Derived] Ji L, Onishi Y, Ahn CW, Agarwal P, Chou CW, Haber H, Guerrettaz K, Boardman MK. Efficacy and safety of exenatide once-weekly vs exenatide twice-daily in Asian patients with type 2 diabetes mellitus. J Diabetes Investig. 2013 Jan 29;4(1):53-61. doi: 10.1111/j.2040-1124.2012.00238.x. Epub 2012 Sep 14. PMID 24843631

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide Once Weekly: Subcutaneous injection of 2 mg exenatide, once a week
- Exenatide Twice Daily: Subcutaneous injection of exenatide, twice a day (5 mcg exenatide per dose for first 4 weeks, then 10 mcg exenatide per dose for 22 weeks)
Period: Overall Study
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Started | 346 | 345
Intent to Treat (ITT) | 340 | 338
Completed | 307 | 266
Not Completed | 39 | 79
Not completed — Adverse Event | 15 | 36
Not completed — Physician Decision | 2 | 4
Not completed — Protocol Violation | 9 | 18
Not completed — Withdrawal by Subject | 5 | 12
Not completed — Lost to follow up | 0 | 2
Not completed — Entry Criteria Not Met | 1 | 0
Not completed — Sponsor Decision | 5 | 5
Not completed — Lack of Efficacy-Loss of Glucose Control | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily | Total
Number analyzed (Participants) | 340 | 338 | 678
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 275 | 274 | 549
  >=65 years | 65 | 64 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (10.59) | 56.2 (9.99) | 55.8 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 154 | 311
  Male | 183 | 184 | 367
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of total hemoglobin] | 8.7 (1.04) | 8.7 (1.03) | 8.7 (1.03)
Weight [Mean (Standard Deviation); unit: kg] | 69.6 (12.44) | 70.4 (12.09) | 70.0 (12.26)
Background Oral Antidiabetic Agent (OAD) [Number; unit: participants]
  Metformin (MET) | 62 | 60 | 122
  MET+Sulfonylurea (SU) | 210 | 216 | 426
  MET+SU+Thiazolidinedione (TZD) | 6 | 10 | 16
  MET+TZD | 12 | 9 | 21
  SU | 30 | 29 | 59
  SU+TZD | 18 | 12 | 30
  TZD | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 26.
Description: Change in HbA1c from baseline to Week 26.
Time Frame: Baseline, Week 26
Population: ITT Population: Randomized patients received at least one dose of study drug. Only patients with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis.
Measure: Least Squares Mean (Standard Error); unit: percentage of total hemoglobin
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 307 | 263
percentage of total hemoglobin | -1.43 (0.07) | -1.12 (0.07)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; MMRM analysis of covariance (ANCOVA) model includes treatment, baseline HbA1c, country, background OAD, week of visit, and treatment-by-week interaction as fixed effects; and patient and error as random effects. Power: 306 patients per treatment group provides approximately 98% power to detect a true difference between treatments of 0.4% in change in HbA1c from baseline with a 2-sided t test at a significance level of 0.05, assuming a common standard deviation of 1.2%; Test type: Non-Inferiority or Equivalence — Superiority of exenatide once weekly to exenatide twice daily concluded if upper limit of the 2-sided 95% confidence interval for treatment difference is <0; noninferiority concluded if upper limit is <0.4%; p < .001, Mixed Models Analysis; Least Squares Mean Difference = -0.31, 95% CI 2-sided [-0.49 to -0.14], Standard Error of Mean 0.09

2. Secondary Outcome: Percentage of Patients Achieving HbA1c Targets <=7% at Week 26
Description: Percentage of patients achieving HbA1c <=7% at Week 26 (for patients with HbA1c >7% at baseline).
Time Frame: Baseline, Week 26
Population: ITT Population. Only patients with baseline HbA1c > target were included in calculation. Only patients with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis. Missing data at endpoint was imputed using last observation carried forward (LOCF) approach.
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 332 | 333
percentage of patients | 46.7 | 35.7
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Percentage of patients achieving HbA1c target <=7% at Week 26 were compared between treatments using a Cochran-Mantel-Haenszel (CMH) test, in which country and background OAD served as the stratification factors; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percentage of Patients Achieving HbA1c Targets <=6.5% at Week 26
Description: Percentage of patients achieving HbA1c <=6.5% at Week 26 (for patients with HbA1c >6.5% at baseline).
Time Frame: Baseline, Week 26
Population: ITT Population. Only patients with baseline HbA1c > target were included in calculation. Only patients with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis. Missing data at endpoint was imputed using LOCF approach.
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 338 | 335
percentage of patients | 26.0 | 15.5
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Percentage of patients achieving HbA1c target <=6.5% at Week 26 were compared between treatments using a CMH test, in which country and background OAD served as the stratification factors; Test type: Superiority or Other; p < .001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Change in Fasting Serum Glucose (FSG) From Baseline to Week 26
Description: Change in FSG from baseline to Week 26.
Time Frame: Baseline, Week 26
Population: ITT Population. Only patients with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 307 | 274
mg/dL | -40.57 (2.36) | -23.90 (2.45)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; MMRM ANCOVA model includes treatment, baseline FSG, country, background OAD, week of visit, and treatment-by-week interaction as fixed effects; and patient and error as random effects; Test type: Superiority or Other; p < .001, Mixed Models Analysis; Least Squares Mean Difference = -16.67, 95% CI 2-sided [-22.50 to -10.83], Standard Error of Mean 2.97

5. Secondary Outcome: Change in Body Weight (BW) From Baseline to Week 26
Description: Change in BW from baseline to Week 26.
Time Frame: Baseline, Week 26
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 309 | 265
kg | -1.63 (0.16) | -2.45 (0.16)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; MMRM ANCOVA model includes treatment, baseline BW, country, background OAD, week of visit, and treatment-by-week interaction as fixed effects; and patient and error as random effects; Test type: Superiority or Other; p < .001, Mixed Models Analysis; Least Squares Mean Difference = 0.82, 95% CI 2-sided [0.39 to 1.25], Standard Error of Mean 0.22

6. Secondary Outcome: Change in Total Cholesterol (TC) From Baseline to Week 26
Description: Change in TC from baseline to Week 26.
Time Frame: Baseline, Week 26
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 309 | 277
mg/dL | -9.41 (1.96) | -8.10 (2.04)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; MMRM ANCOVA model includes treatment, baseline TC, country, background OAD, week of visit, and treatment-by-week interaction as fixed effects; and patient and error as random effects; Test type: Superiority or Other; p = 0.609, Mixed Models Analysis; Least Squares Mean Difference = -1.31, 95% CI 2-sided [-6.33 to 3.71], Standard Error of Mean 2.56

7. Secondary Outcome: Change in High-Density Lipoprotein (HDL) From Baseline to Week 26
Description: Change in HDL from baseline to Week 26.
Time Frame: Baseline, Week 26
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 309 | 277
mg/dL | -0.11 (0.41) | -0.48 (0.43)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; MMRM ANCOVA model includes treatment, baseline HDL, country, background OAD, week of visit, and treatment-by-week interaction as fixed effects; and patient and error as random effects; Test type: Superiority or Other; p = 0.476, Mixed Models Analysis; Least Squares Mean Difference = 0.37, 95% CI 2-sided [-0.65 to 1.38], Standard Error of Mean 0.52

8. Secondary Outcome: Ratio of Triglycerides (TG) at Week 26 to Baseline
Description: Ratio of TG (measured in mg/dL) at Week 26 to baseline. Log(Post-baseline TG) - log(Baseline TG); change from baseline to Week 26 is presented as ratio of Week 26 to baseline.
Time Frame: Baseline, Week 26
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 309 | 277
ratio | 0.97 (0.02) | 0.97 (0.03)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; TG data were logarithm-transformed and the change at Week 26 to baseline, expressed as the ratio, was analyzed using a MMRM ANCOVA model with treatment, baseline TG, country, background OAD, week of visit, and treatment-by-week interaction as fixed effects; and patient and error as random effects; Test type: Superiority or Other; p = 0.807, Mixed Models Analysis; Geometic Least Squares Mean Ratio = 0.99, 95% CI 2-sided [0.93 to 1.06], Standard Error of Mean 0.03

9. Secondary Outcome: Change in Blood Pressure From Baseline to Week 26
Description: Change in systolic blood pressure and diastolic blood pressure from baseline to Week 26.
Time Frame: Baseline, Week 26
Population: ITT Population. Only patients with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis. Missing data at endpoint was not imputed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 337 | 335
mmHg
  Systolic Blood Pressure | -5.33 (15.99) | -5.22 (16.23)
  Diastolic Blood Pressure | -1.47 (9.52) | -2.24 (9.56)

10. Secondary Outcome: Assessment of Event Rate of Treatment-emergent Hypoglycemic Events
Description: Major hypoglycemia: any episode with symptoms consistent with hypoglycemia that resulted in loss of consciousness or seizure with prompt recovery in response to administration of glucagon or glucose OR documented hypoglycemia (blood glucose <3.0 mmol/L [54 mg/dL]) and required the assistance of another person. Minor hypoglycemia: any sign or symptom associated with hypoglycemia that is either self-treated by the patient or resolves on its own AND has a concurrent finger stick blood glucose <3.0 mmol/L (54 mg/dL) and not classified as major hypoglycemia. Event rate per subject year was calculated for each subject: (number of events observed from a subject/exposure from a subject)*365.25 where exposure = last post-baseline visit date - baseline visit date. Mean and Standard Error were then derived from ITT.
Time Frame: Baseline to Week 26
Population: ITT Population.
Measure: Mean (Standard Error); unit: events per subject-year
Groups:
- Exenatide Once Weekly With SU Use at Screening: Subcutaneous injection of 2 mg exenatide, once a week and with SU use at Screening
- Exenatide Twice Daily With SU Use at Screening: Subcutaneous injection of exenatide, twice a day (5 mcg exenatide per dose for first 4 weeks, then 10 mcg exenatide per dose for 22 weeks) and with SU use at Screening
- Exenatide Once Weekly Without SU Use at Screening: Subcutaneous injection of 2 mg exenatide, once a week and without SU use at Screening
- Exenatide Twice Daily Without SU Use at Screening: Subcutaneous injection of exenatide, twice a day (5 mcg exenatide per dose for first 4 weeks, then 10 mcg exenatide per dose for 22 weeks) and without SU use at Screening
Arm/Group | Exenatide Once Weekly With SU Use at Screening | Exenatide Twice Daily With SU Use at Screening | Exenatide Once Weekly Without SU Use at Screening | Exenatide Twice Daily Without SU Use at Screening
Number analyzed (Participants) | 264 | 267 | 76 | 71
events per subject-year
  Major Hypoglycemia | 0.00 (0.000) | 0.01 (0.007) | 0.00 (0.000) | 0.00 (0.000)
  Minor Hypoglycemia | 0.24 (0.069) | 0.59 (0.180) | 0.03 (0.027) | 0.11 (0.113)

ADVERSE EVENTS:
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Serious Adverse Events (participants affected / at risk) | 13/340 | 8/338
Other Adverse Events (participants affected / at risk) | 131/340 | 150/338
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (N=340) | Exenatide Twice Daily (N=338)
Cerebral infarction (Nervous system disorders) | 2 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Blood calcitonin increased (Investigations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Cerebral artery occlusion (Nervous system disorders) | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Diplegia (Nervous system disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Pneumonia haemophilus (Infections and infestations) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Transient global amnesia (Nervous system disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (N=340) | Exenatide Twice Daily (N=338)
Injection site induration (General disorders) | 33 | 2
Diarrhoea (Gastrointestinal disorders) | 32 | 27
Nausea (Gastrointestinal disorders) | 32 | 73
Vomiting (Gastrointestinal disorders) | 27 | 39
Dyslipidaemia (Metabolism and nutrition disorders) | 21 | 23
Constipation (Gastrointestinal disorders) | 20 | 24
Injection site nodule (General disorders) | 18 | 0
Injection site pruritus (General disorders) | 18 | 9
Decreased appetite (Metabolism and nutrition disorders) | 15 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days